CLINICAL TRIAL: NCT02862665
Title: Effect of Perioperative Iron Isomaltoside 1000 Administration on Transfusion Requirements in Patients Undergoing Complex Valvular Heart Surgery: a Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4-2016-0502
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Complex Valvular Heart Surgery
MeSH Terms: interventions — iron isomaltoside 1000; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV iron (Experimental): The patients will receive iron isomaltoside 1000 (Monofer®) as an i.v. infusion of 1000 mg (diluted with normal saline, 10 mg/ml) twice; 3 days before surgery and 3 days after surgery. They will receive iron isomaltoside 1000 (Monofer®) 1000 mg over 15 min.
  Interventions: Drug: iron isomaltoside 1000 (Monofer®)
- Control (Placebo Comparator): The patients will receive normal saline 100 ml as an i.v. infusion twice; 3 days before surgery and 3 days after surgery. They will receive normal saline 100 ml over 15 min.
  Interventions: Drug: normal saline 100 ml

INTERVENTIONS:
Drug: iron isomaltoside 1000 (Monofer®) — The patients will receive iron isomaltoside 1000 (Monofer®) as an i.v. infusion of 1000 mg (diluted with normal saline, 10 mg/ml) twice; 3 days before surgery and 3 days after surgery. They will receive iron isomaltoside 1000 (Monofer®) 1000 mg over 15 min.
  Arms: IV iron
Drug: normal saline 100 ml — The patients will receive normal saline 100 ml as an i.v. infusion twice; 3 days before surgery and 3 days after surgery. They will receive normal saline 100 ml over 15 min.
  Arms: Control

SUMMARY:
In complex cardiac surgery with prolonged cardiopulmonary bypass, allogeneic blood products transfusions are often necessary to control intraoperative and postoperative bleeding. Furthermore, approximately 50% of all patients undergoing cardiac surgery are anemic before surgery, and patients with normal hemoglobin level may become anemic during and/or after surgery. Perioperative transfusion carries risks far beyond transmission of infection and has been demonstrated to be associated with adverse outcomes related to postoperative pulmonary complications, decreased renal function and increased mortality. Thus, the important of blood conservation stratigies to minimize transfusion is being increasingly emphasized. In recent trial by Johansson and colleagues, they concluded that the perioperative administration of intravenous iron isomaltoside 1000 increased the hemoglobin level and prevented anemia 4 weeks after cardiac surgery. Therefore, perioperative iron isomaltoside 1000 administration among the patients undergoing complex valvular heart surgery could reduce not only the perioperative allogeneic transfusion but also the incidence of postoperative adverse events. The aim of this study is to examine the effect of perioperative iron isomaltoside 1000 administration on transfusion requirements in patients undergoing complex valvular heart surgery.

ELIGIBILITY:
Inclusion Criteria:

1. the patients undergoing redo cardiac surgery or complex valvular heart surgery with cardiopulmonary bypass
2. tha age ≥19 yrs old.
3. the patients who are willing to provide written informed consent

Exclusion Criteria:

1. having preoperative anemia (Hb <9 g/dl for women, Hb <10 g/dl for men)
2. preoperative erythropoietin treatment within four weeks before surgery
3. redo cardiac operation due to preoperative paravalvular leakage
4. known hypersensitivity to any excipients in the investigational drug products
5. aplastic anemia
6. the patients who stay more than 48 hours in the intensive care unit preoperatively due to heart failure or other major complication

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-05-07 (Actual)

PRIMARY OUTCOMES:
the proportion of patients who need blood transfusion | patients will be followed for the duration of hospital stay, an expected average of 10 days after surgery
  Investigator will assess the number of patients in each group who will need blood transfusion during hospital stays, and evaluate the effect of iron isomaltoside 1000 (Monofer®) on perioperative blood transfusion.

SECONDARY OUTCOMES:
the proportion of patients who will experience postoperative adverse events | within the first 20 days after surgery. (plus or minus 3 days)
  Investigator will assess the number of patients in each group who will experience postoperative adverse events (death, atrial fibrillation, reoperation, wound infection, acute kidney injury, permanent stroke, prolonged mechanical ventilation or postoperative myocardial infarction) within the first 20 days after surgery, and evaluate the effect of iron isomaltoside 1000 (Monofer®) on the occurrence of any postoperative adverse events.
the plasma hepcidin concentrations of patients | before the investigational drug i.v. infusion; 3 days before surgery and 3 days after surgery
  Investigator will assess the plasma hepcidin concentrations before the investigational drug i.v. infusion; 3 days before surgery and 3 days after surgery, and evaluate the association between the plasma hepcidin concentrations and the effect of iron isomaltoside 1000 (Monofer®) or the occurrence of any postoperative adverse events.
the plasma EPO (erythropoietin) concentrations of patients | before the investigational drug i.v. infusion; 3 days before surgery and 3 days after surgery
  Investigator will assess the plasma EPO concentrations before the investigational drug i.v. infusion; 3 days before surgery and 3 days after surgery, and evaluate the association between the plasma EPO concentrations and the effect of iron isomaltoside 1000 (Monofer®) or the occurrence of any postoperative adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Thoracic and Cardiovascular Surgery, Cardiovascular Research Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee SH, Shim JK, Soh S, Song JW, Chang BC, Lee S, Kwak YL. The effect of perioperative intravenously administered iron isomaltoside 1000 (Monofer(R)) on transfusion requirements for patients undergoing complex valvular heart surgery: study protocol for a randomized controlled trial. Trials. 2018 Jul 4;19(1):350. doi: 10.1186/s13063-018-2545-3. PMID 29973224